CLINICAL TRIAL: NCT02878317
Title: Association of Advanced Glycation End-product Accumulation and Adverse Outcomes in Peritoneal Dialysis and Haemodialysis Patients and the Impact of a Dietetic Intervention on Skin Autofluorescence
Brief Title: Skin Autofluorescence as a Risk Marker in People Receiving Dialysis.
Acronym: AGED
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16050
Record Dates: First submitted 2016-08-05; First posted 2016-08-25 (Estimated); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Disease
Keywords: Glycosylation End Products, Advanced; Skin autofluorescence; Renal Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study 2 - Non randomised proof of principle study: Malnourished participants received individualized nutritional advice and support formulated and delivered by experienced dietitians consisting of food fortification recommendations and oral nutritional supplementation aiming to achieve estimated nutritional requirements (i.e. energy [30-35 kcal/kg/day] and protein intake [1.1-1.2 g/kg/day]). Food fortification involved enhancing the energy and protein content of meals and snacks without increasing the portion sizes of foods. Advice was individualized according to patient needs and food preferences. Oral nutritional supplements included Fortisip Compact (2.4 kcal/ml), Fortisip (1.5 kcal/ml) and Fortijuice (1.5 kcal/ml), as well as Renapro® shot and Fresubin® 5kcal Shot.
- Historical control group from Study 1: Participants on dialysis with malnutrition taken from Study 1, who were seen by their usual dietitian once a month and received standard nutritional counselling.

SUMMARY:
The purpose of the present study is to investigate the association between the accumulation of advanced glycation end-products (AGE) and adverse outcomes (e.g. death) in people receiving haemodialysis and peritoneal dialysis based in Royal Derby Hospital, as well as the impact of a dietetic intervention on AGE accumulation. AGE will be measured non-invasively in the skin using a technique called skin autofluorescence (SAF).

The present study will be conducted in two parts:

Study 1: this will be a prospective study where participants will be followed-up for up to five years. The research team will measure the accumulation of AGE in the skin using a quick (less than five minutes) and painless technique called SAF. This involves placing the forearm on a piece of equipment that shines a light on the skin and measures the amount of light that is reflected back. Participants will be asked to complete nutritional and quality of life questionnaires, measurements of weight, height, arm circumference and skinfold thickness (i.e. anthropometry), simple eyesight tests and blood tests.

Study 2: observational non-randomized proof of principle study where malnourished dialysis participants will receive a dietitian supervised intensive nutritional support. Participants will be followed-up for 2 years and will receive precise oral and written instructions on how to comply with the intervention. Blood and eyesight tests, SAF measurements, anthropometry and nutritional and quality of life assessments will be conducted.

In Studies 1 and 2, approximately two teaspoons of blood will be collected to measure AGE levels and do some additional blood tests to help us investigate the effects of AGEs on the body. If the participants agree, the investigators will also store some of the blood for future research.

DETAILED DESCRIPTION:
STUDY BACKGROUND

Chronic kidney disease (CKD) is a global public health problem and is associated with multiple adverse outcomes including reduced survival, especially in people requiring renal replacement therapy (peritoneal dialysis (PD), haemodialysis [HD] and transplantation). Multiple risk factors lead to the development and/or progression of CKD, such as obesity, hyperlipidaemia, glomerulonephritis, intercurrent infections, smoking, type 2 diabetes and hypertension, the two latter being considered as leading causes of CKD worldwide.

People on dialysis develop a variety of complications/abnormalities as a result of loss of endocrine or exocrine function of the kidneys, including anaemia, metabolic acidosis, bone and mineral disorders, fluid overload, hypertension, electrolyte disturbances and dyslipidaemia. In recent years, inflammation, oxidative stress and endothelial dysfunction (other common abnormalities in people on dialysis) have become areas of interest because of their strong relationship with higher rates of cardiovascular morbidity and mortality in people on dialysis.

Advanced glycation end-products (AGE) are uremic toxins that are markedly increased in people on dialysis. Formation of AGE starts with a non-enzymatic reaction between proteins and glucose molecules called the Maillard reaction; however, AGE are also formed more rapidly during oxidative stress with the subsequent formation of reactive carbonyl compounds like methyl glyoxal. At this point, AGE synthesis is irreversible and AGE will cross-link with tissue proteins; it seems that collagen in the skin and vascular basement membranes are especially susceptible to AGE accumulation and subsequent injury. AGE also interact with specific AGE receptors that will lead to the activation of systemic inflammation by increasing the release of cytokines and, consequently, exacerbate tissue damage. Importantly, AGE are also formed in food during cooking with dry heat at high temperatures such as in frying, grilling or roasting and about 10% of the ingested AGE is absorbed.

Skin autofluorescence (SAF) is a relatively new technique that measures the skin accumulation of AGE. It is a non-invasive, operator independent, quick (less than 5 minutes) and easy to perform technique that utilizes the fluorescent properties of AGE, like the extensively used collagen linked fluorescence (CLF) method, and has been validated with specific AGE measurements and CLF in skin biopsies. It has been reported that SAF is strongly correlated with overall and cardiovascular mortality in people with diabetes and undergoing HD. Several factors have been associated with higher SAF values in people on dialysis in cross-sectional studies, for instance, chronological age in both dialysis modalities, glucose exposure from peritoneal dialysis fluid and dialysis vintage only in people on PD and presence of diabetes in people on HD.

AGE accumulation is postulated as the one of the modulating factors that drives visual disorders; the increased accumulation secondary to hyperglycaemia in diabetes is thought to cause vascular basement membrane thickening and destruction of pericytes from the retinal capillary bed in diabetic retinopathy. The accumulation of AGE has also been reported to be a mechanism in the deterioration in visual acuity associated with increasing age. Separately, the accumulation of AGE in other metabolic diseases (e.g. end stage kidney disease [ESKD]) has been found to cause nerve and eye dysfunction. Ocular abnormalities and therefore visual disturbances are reported in people with ESKD but the mechanism for this has not been fully explored or understood. In animal studies, AGE accumulation is seen in the lens, cornea and vitreous humour. In humans, systemic AGE levels and visual acuity scoring have not been previously investigated.

Because of the adverse outcomes strongly associated with higher levels of SAF, several options focused on reducing the accumulation of AGE have been proposed. One of these promising interventions is the reduction of dietary AGE; it has been suggested that cooking techniques that avoid very high temperatures such as poaching, steaming, stewing and boiling can significantly reduce the AGE content of food when compared to frying, broiling, grilling and roasting; nevertheless, most of the evidence regarding dietary modifications to reduce exogenous AGE is of low quality and therefore further studies are required.

Nevertheless, analysis of baseline data from Study 1 has identified strong associations between higher SAF and malnutrition whereas no correlations were observed between higher SAF and high dietary AGE intake. Correction of malnutrition may therefore represent a more important dietary intervention to reduce accumulation of AGE in people receiving dialysis. We further reasoned that placing people with malnutrition on a restrictive diet may worsen their malnutrition and we have therefore adapted our original research plan to include an observational study to assess the impact of correcting malnutrition on SAF by providing a dietitian supervised nutritional support intervention, which essentially involves the usual/standard dietetic care/advice provided by the NHS with some additional supervision, follow-up and approved dietary supplements (also provided by the NHS), rather than a randomised trial of dietary AGE restriction.

The results from the present project will benefit people on dialysis because they may demonstrate that the correction of malnutrition decreases the SAF levels in this population. Published observational studies suggest that reduction of SAF levels will in turn be associated with a reduction in the high morbidity and mortality rates associated with chronic dialysis and, consequently, healthcare costs. Improved survival and reduced comorbidity would also be expected to improve the quality of life of people on dialysis.

DURATION OF THE STUDY

Study 1:

Participant recruitment will begin on September 2016 with an anticipated recruitment period of 12 months. Therefore, all baseline data and measurements will be collected and performed between September 2016 and September 2017. Once recruited, all participants will be followed-up for up to five years; consequently, it is expected that the study will be completed by September 2022.

Study 2:

Participant recruitment will begin in December 2017 with an anticipated recruitment period of 6 months. Therefore, all baseline data and measurements will be collected and performed between December 2017 and June 2018. Once recruited, all participants will be followed-up for 24 months; consequently, it is expected that the study will be completed by June 2020.

RECRUITMENT

Potential participants on HD and PD will be recruited from the Renal Unit of the Department of Nephrology at the Royal Derby Hospital. The initial details of the study and participant information sheet will be provided by the usual care team (which may include the researcher). Participants will then be given at least 24 hours to consider whether they wish to participate, as well as ask any questions about the study, before being re-contacted by the investigators.

INFORMED CONSENT

The process for obtaining participant informed consent will be in accordance with the Research Ethics Committee (REC) guidance, Good Clinical Practice (GCP) and any other regulatory requirements that might be introduced.

All participants will provide written informed consent. The Informed Consent Form will be signed and dated by the participant before they enter the study. The Investigator will explain the details of the study and provide a Participant Information Sheet, ensuring that the participant has sufficient time to consider participating or not. The Investigator will answer any questions that the participant has concerning study participation.

STATISTICS

To compare baseline versus final evaluations, Wilcoxon test or paired t-test will be used in the case of dimensional variables, and McNemar test in the case of categorical variables. Intergroup comparisons will be performed using Mann Whitney test or Student t test for continuous variables and χ2 test or Fisher's exact test for categorical variables. To determine the significance and strength of associations, Pearson's correlation coefficient will be used for analyses of associations between continuous variables and Spearman rank for nonparametric variables. Linear regression analysis will be used to identify determinants of AGE accumulation. Cox proportional hazards models will be used to investigate the prognostic value of the accumulation of AGE for predicting mortality. A p-value less than or equal to 0.05 will be considered to have statistical significance.

Sample size calculation of Study 1 was performed by using the software nQuery Advisor v.6.0.

Sample size Study 1:

The primary outcome for sample size determination is one-year survival in relation to increased SAF levels in people on HD and PD. With a power of 80%, a two-sided alpha of 5% and an expected hazard ratio of 3.5 and 2.0 in people on PD and HD, respectively, 100 HD and 40 PD participants will be needed.

Sample size Study 2 Since this is a proof of principle study, it would be reasonable to include 40 dialysis participants (either HD or PD).

ETHICS COMMITTEE AND REGULATORY APPROVALS

The study will not be initiated before the protocol, informed consent forms and participant information sheets have received approval / favourable opinion from the REC, and the respective NHS Research & Development (R&D) department.

PROCEDURES FOR MISSING DATA AND ADVERSE EVENTS

All SAF measurements, biochemistry, nutritional and quality of life assessments for Study 1 and 2 will be used in the statistical analysis, including data from participants who did not complete the entire study protocol.

The occurrence of an adverse event as a result of participation within this study is not expected and as such no adverse event data will be collected.

QUALITY ASSURANCE & AUDIT

Study conduct may be subject to systems audit of the Trial Master File for inclusion of essential documents; permissions to conduct the study; Trial Delegation Log; CVs of study staff and training received; local document control procedures; consent procedures and recruitment logs; adherence to procedures defined in the protocol (e.g. inclusion / exclusion criteria, correct randomisation, timeliness of visits); AE recording and reporting; accountability of study materials and equipment calibration logs.

Monitoring of study data shall include confirmation of informed consent; source data verification; data storage and data transfer procedures; local quality control checks and procedures, back-up and disaster recovery of any local databases and validation of data manipulation.

Entries on Case Report Forms (CRFs) will be verified by inspection against the source data. A sample of CRFs (10% or as per the study risk assessment) will be checked on a regular basis for verification of all entries made. In addition the subsequent capture of the data on the study database will be checked. Where corrections are required these will carry a full audit trail and justification.

Study data and evidence of monitoring and systems audits will be made available for inspection by REC as required.

ELIGIBILITY:
Inclusion Criteria:

Haemodialysis cohort:

* Three dialysis sessions per week for 4 hours.
* Dialysis with biocompatible membranes.
* Able to give informed consent.

Peritoneal Dialysis cohort:

* Dialysis with lactate/bicarbonate-buffered solutions with different glucose concentrations as prescribed for routine clinical care.
* Able to give informed consent.

Exclusion Criteria:

* Does not wish to participate.
* Renal transplant.
* Pregnancy or breast feeding or intending pregnancy.
* Expected survival less than one year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing HD and PD treatment.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Taal, Doctor, Study Director — University Hospitals of Derby and Burton NHS Foundation Trust
Locations (1):
- Derby Hospitals NHS Foundation Trust, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arsov S, Graaff R, van Oeveren W, Stegmayr B, Sikole A, Rakhorst G, Smit AJ. Advanced glycation end-products and skin autofluorescence in end-stage renal disease: a review. Clin Chem Lab Med. 2014 Jan 1;52(1):11-20. doi: 10.1515/cclm-2012-0832. PMID 23612551
- [Background] Darlene, A., Dartt Reza, D. and D'Amore, P. (2011) Immunology, inflammation and diseases of the eye. Elsevier Press: pp. 287-288.
- [Background] Graaff R, Arsov S, Ramsauer B, Koetsier M, Sundvall N, Engels GE, Sikole A, Lundberg L, Rakhorst G, Stegmayr B. Skin and plasma autofluorescence during hemodialysis: a pilot study. Artif Organs. 2014 Jun;38(6):515-8. doi: 10.1111/aor.12205. Epub 2013 Oct 29. PMID 24164288
- [Background] Hartog JW, Voors AA, Schalkwijk CG, Scheijen J, Smilde TD, Damman K, Bakker SJ, Smit AJ, van Veldhuisen DJ. Clinical and prognostic value of advanced glycation end-products in chronic heart failure. Eur Heart J. 2007 Dec;28(23):2879-85. doi: 10.1093/eurheartj/ehm486. Epub 2007 Nov 5. PMID 17986469
- [Background] Ishibashi T, Murata T, Hangai M, Nagai R, Horiuchi S, Lopez PF, Hinton DR, Ryan SJ. Advanced glycation end products in age-related macular degeneration. Arch Ophthalmol. 1998 Dec;116(12):1629-32. doi: 10.1001/archopht.116.12.1629. PMID 9869793
- [Background] Junaid Nazar CM, Kindratt TB, Ahmad SM, Ahmed M, Anderson J. Barriers to the successful practice of chronic kidney diseases at the primary health care level; a systematic review. J Renal Inj Prev. 2014 Jul 1;3(3):61-7. doi: 10.12861/jrip.2014.20. eCollection 2014. PMID 25340171
- [Background] Kandarakis SA, Piperi C, Topouzis F, Papavassiliou AG. Emerging role of advanced glycation-end products (AGEs) in the pathobiology of eye diseases. Prog Retin Eye Res. 2014 Sep;42:85-102. doi: 10.1016/j.preteyeres.2014.05.002. Epub 2014 Jun 4. PMID 24905859
- [Background] Kellow NJ, Savige GS. Dietary advanced glycation end-product restriction for the attenuation of insulin resistance, oxidative stress and endothelial dysfunction: a systematic review. Eur J Clin Nutr. 2013 Mar;67(3):239-48. doi: 10.1038/ejcn.2012.220. Epub 2013 Jan 30. PMID 23361161
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD Work Group (2013). KDIGO 2012 Clinical practice guideline for the evaluation and management of chronic kidney disease. Kidney Int 4(Suppl. 3): pp. 1-150.
- [Background] Kimura H, Tanaka K, Kanno M, Watanabe K, Hayashi Y, Asahi K, Suzuki H, Sato K, Sakaue M, Terawaki H, Nakayama M, Miyata T, Watanabe T. Skin autofluorescence predicts cardiovascular mortality in patients on chronic hemodialysis. Ther Apher Dial. 2014 Oct;18(5):461-7. doi: 10.1111/1744-9987.12160. Epub 2014 Jan 24. PMID 24456287
- [Background] McIntyre NJ, Chesterton LJ, John SG, Jefferies HJ, Burton JO, Taal MW, Fluck RJ, McIntyre CW. Tissue-advanced glycation end product concentration in dialysis patients. Clin J Am Soc Nephrol. 2010 Jan;5(1):51-5. doi: 10.2215/CJN.05350709. Epub 2009 Nov 5. PMID 19965551
- [Background] Nongnuch A, Davenport A. The effect of vegetarian diet on skin autofluorescence measurements in haemodialysis patients. Br J Nutr. 2015 Apr 14;113(7):1040-3. doi: 10.1017/S0007114515000379. Epub 2015 Mar 12. PMID 25761438
- [Background] Oleniuc M, Schiller A, Secara I, Onofriescu M, Hogas S, Apetrii M, Siriopol D, Covic A. Evaluation of advanced glycation end products accumulation, using skin autofluorescence, in CKD and dialysis patients. Int Urol Nephrol. 2012 Oct;44(5):1441-9. doi: 10.1007/s11255-011-0097-5. Epub 2011 Dec 10. PMID 22160646
- [Background] Siriopol D, Hogas S, Veisa G, Mititiuc I, Volovat C, Apetrii M, Onofriescu M, Busila I, Oleniuc M, Covic A. Tissue advanced glycation end products (AGEs), measured by skin autofluorescence, predict mortality in peritoneal dialysis. Int Urol Nephrol. 2015 Mar;47(3):563-9. doi: 10.1007/s11255-014-0870-3. Epub 2014 Nov 26. PMID 25425437
- [Background] Smit AJ, Gerrits EG. Skin autofluorescence as a measure of advanced glycation endproduct deposition: a novel risk marker in chronic kidney disease. Curr Opin Nephrol Hypertens. 2010 Nov;19(6):527-33. doi: 10.1097/MNH.0b013e32833e9259. PMID 20844429
- [Background] Uribarri J, Woodruff S, Goodman S, Cai W, Chen X, Pyzik R, Yong A, Striker GE, Vlassara H. Advanced glycation end products in foods and a practical guide to their reduction in the diet. J Am Diet Assoc. 2010 Jun;110(6):911-16.e12. doi: 10.1016/j.jada.2010.03.018. PMID 20497781
- [Background] Singh VP, Bali A, Singh N, Jaggi AS. Advanced glycation end products and diabetic complications. Korean J Physiol Pharmacol. 2014 Feb;18(1):1-14. doi: 10.4196/kjpp.2014.18.1.1. Epub 2014 Feb 13. PMID 24634591
- [Background] Zhang QL, Rothenbacher D. Prevalence of chronic kidney disease in population-based studies: systematic review. BMC Public Health. 2008 Apr 11;8:117. doi: 10.1186/1471-2458-8-117. PMID 18405348
- [Background] Wright M, Jones C. Renal Association Clinical Practice Guideline on nutrition in CKD. Nephron Clin Pract. 2011;118 Suppl 1:c153-64. doi: 10.1159/000328067. Epub 2011 May 6. No abstract available. PMID 21555894

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study 1:
  Participant recruitment began in September 2016. All baseline data and measurements were collected and performed between September 2016 and August 2017. Once recruited, all participants were followed-up for up to five years.
  Study 2:
  Participant recruitment began in December 2017. All baseline data and measurements were collected and performed between December 2017 and June 2018. Once recruited, all participants were followed-up for up to 24 months.
Groups:
- Study 2 - Non Randomised Proof of Principle Study: Malnourished participants received individualized nutritional advice and support formulated and delivered by experienced dietitians consisting of food fortification recommendations and oral nutritional supplementation aiming to achieve estimated nutritional requirements (i.e. energy [30-35 kcal/kg/day] and protein intake [1.1-1.2 g/kg/day]). Food fortification involved enhancing the energy and protein content of meals and snacks without increasing the portion sizes of foods. Advice was individualized according to patient needs and food preferences. Oral nutritional supplements included Fortisip Compact (2.4 kcal/ml), Fortisip (1.5 kcal/ml) and Fortijuice (1.5 kcal/ml) (Nutricia Advanced Medical Nutrition®, Wiltshire, United Kingdom), as well as Renapro® shot (Stanningly Pharma, BioCity, Pennyfoot Street, Nottingham, United Kingdom) and Fresubin® 5kcal Shot (Fresenius Kabi Ireland, Balbriggan, Dublin, Ireland).
  Participants received precise oral and written instructions on how and when to take the supplements and how to follow the food fortification advice provided. Participants were closely monitored by the dietitian at least once a week to encourage adherence to nutritional advice, and 24-hour dietary recalls were also conducted to ensure compliance with the advice provided. Each participant was also reviewed quarterly with the clinical lead renal dietitian in order to modify the dietetic advice, if required.
Period: Overall Study
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Started | 32 | 49
Completed | 28 | 49
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Study 2: Baseline data is for the 28 malnourished participants who completed 6 months of follow-up
- Historical Control Group - Study 1: A historical control group of malnourished persons on dialysis (n=41 haemodialysis and 8 peritoneal dialysis) taken from Study 1 (observational study).
- Total: Total of all reporting groups
Arm/Group | Study 2 | Historical Control Group - Study 1 | Total
Number analyzed (Participants) | 28 | 49 | 77
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65 [56 to 74] | 63 [53 to 75] | 64 [54.5 to 74.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 26 | 40
  Male | 14 | 23 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 43 | 67
  More than one race | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Serum albumin [Median (Inter-Quartile Range); unit: g/L] | 30.0 [26.0 to 33.0] | 32.0 [27.0 to 34.0] | 31.0 [26.5 to 33.5]
Dietary AGE intake [Median (Inter-Quartile Range); unit: Kilounits/day] — Quantification of advanced glycation end-products (AGEs) in food was determined with a food frequency questionnaire previously validated in a diabetic population. Dietary AGE intake was reported in kilounits/day (kU/day).
  Kilounits/day | 13823 [10840 to 20441] | 11940 [8787 to 15833] | 12882 [9814 to 18137]
Energy intake [Median (Inter-Quartile Range); unit: kcal/kg/day] — Information regarding energy intake was obtained from three 24-hour dietary recalls including one dialysis day and one week-end day. Dietary recalls were analysed using the software Dietplan 7 (Forestfield Software Limited,West Sussex, United Kingdom) to calculate the average energy intake. The average daily intake of calories was then calculated in kilocalories and expressed per kilogram of ideal body weight.
  kcal/kg/day | 20.9 [16.6 to 27.3] | 17.9 [13.5 to 21.7] | 19.4 [15.1 to 24.5]
Protein intake [Median (Inter-Quartile Range); unit: g/kg/day] — Information regarding protein intake was obtained from three 24-hour dietary recalls including one dialysis day and one week-end day. Dietary recalls were analysed using the software Dietplan 7 (Forestfield Software Limited,West Sussex, United Kingdom) to calculate the average protein intake. The average daily intake of protein was then calculated in grams, and expressed per kilogram of ideal body weight.
  g/kg/day | 0.7 [0.6 to 1.1] | 0.8 [0.6 to 1.0] | 0.75 [0.6 to 1.05]
Skin autofluorescence [Mean (Standard Deviation); unit: Arbitrary units] — Tissue AGE accumulation as assessed by skin autofluorescence (SAF) was measured with a validated Autofluorescence Reader, version 2.4.3 (AGE Reader SU, DiagnOptics Technologies). The AGE Reader SU directs an ultraviolet excitation light through an illumination window on a skin area of the volar surface of the forearm at 10 cm below the elbow. The AGE Reader SU then measures the emission light using a spectrometer and a 200-mm glass fibre. SAF is calculated by dividing the average emitted light intensity by the average excitation light intensity and expressed as arbitrary units.
  Arbitrary units | 3.8 (0.7) | 3.5 (0.9) | 3.7 (0.8)
Handgrip strength [Median (Inter-Quartile Range); unit: kg] — Handgrip strength (HGS) measurement was conducted within the first hour of haemodialysis treatment or during peritoneal dialysis clinic visits using the Takei 5401 handgrip digital dynamometer (Takei Scientific Instruments Co., Ltd., Tokyo, Japan). HGS was measured in the non-fistula arm or the dominant arm if the participant did not have a fistula. Participants were instructed to apply maximum handgrip pressure and then relaxed. HGS was expressed in kilograms.
  kg | 15.2 [10.4 to 22.3] | 17.3 [12.2 to 25.6] | 16.3 [11.3 to 23.9]

OUTCOME MEASURES:

1. Primary Outcome: Skin Autofluorescence Levels at 6 Months
Description: Skin autolfuorescence (SAF) was measured after 6 months of intensive dietetic advice and nutritional support with a validated Autofluorescence Reader (AGE) Standard Unit (SU), version 2.4.3. The AGE Reader SU directs an ultraviolet excitation light through an illumination window of approximately 1 cm2 on a skin area of the volar surface of the forearm at approximately 10 cm below the elbow. The AGE Reader then measures the amount of emitted light that is reflected back from the skin using a spectrometer and a 200-µm glass fiber. SAF is calculated as the ratio between emission and excitation and is expressed as arbitrary units (AU). Three measurements were conducted and the mean value of these was used for statistical analysis. The reference value of SAF for the age group of 60-70 years is 2.5±0.6 AU.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Arbitrary units
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 49
Arbitrary units | 3.7 (0.7) | 3.8 (1.2)

2. Secondary Outcome: Energy Intake at 6 Months.
Description: Energy (calorie) intake after 6 months of intensive dietetic advice and nutritional support.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Kcal/kg/day
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 49
Kcal/kg/day | 30.1 [24.9 to 35.9] | 18.9 [15.1 to 26.9]

3. Secondary Outcome: Nutritional Status at 6 Months
Description: The 7-point scale Subjective Global Assessment (SGA, gold standard for nutritional status assessment in the dialysis population) was used to evaluate nutritional status at 6 months after intensive dietetic advice and nutritional support. The SGA score ranges from 1-7. Nutritional status can be classified into normal nutritional status (scores of 6 or 7), mild-moderate malnutrition (scores of 3-5), or severe malnutrition (scores of 1 or 2).
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 49
score on a scale | 5.0 [5.0 to 6.0] | 5.0 [3.0 to 7.0]

4. Secondary Outcome: Dietary Advanced Glycation End-products (AGE) Intake at 6 Months
Description: Dietary AGE intake after 6 months of intensive dietetic advice and nutritional support
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: Kilounits/day
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 49
Kilounits/day | 19074 [13372 to 27340] | 14697 [9427 to 19071]

5. Secondary Outcome: Protein Intake at 6 Months.
Description: Protein intake after 6 months of intensive dietetic advice and nutritional support.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: g/kg/day
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 49
g/kg/day | 1.1 [0.8 to 1.2] | 0.8 [0.6 to 1.0]

6. Secondary Outcome: Serum Albumin Levels at 6 Months
Description: Serum albumin levels after 6 months of intensive dietetic advice and nutritional support.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 49
g/L | 31.5 [30.0 to 34.0] | 31.0 [27.0 to 34.5]

7. Secondary Outcome: Handgrip Strength at 6 Months
Description: Handgrip strength after 6 months of intensive dietetic advice and nutritional support.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 49
kg | 16.7 [10.6 to 24.7] | 18.3 [12.4 to 26.3]

8. Other Pre Specified Outcome: Health-related Quality of Life, Short Form-36 Physical Component Score
Description: The Short Form-36 (SF-36) physical component score (PCS) was calculated after 6 months of intensive dietetic advice and nutritional support according to well-defined guidelines as follows: 1) recoding of 10 questions of the SF-36 survey; 2) calculation of raw scores for each of the eight health state domains of the SF-36 survey; 3) transformation of raw scores into a 0-100 scale; 4) standardisation of the transformed scales using a z-score transformation and the means and standard deviations from the general United Kingdom (UK) population; 5) calculation of the PCS by multiplying each scale z-score by their respective physical factor score coefficient and summing the eight products; and 6) the resulting sum is multiplied by 10 and added to 50 to linearly transform the PCS to the T-score metric, which has a mean of 50 and a standard deviation of 10 for the general UK population. A PCS above or below 50 is therefore indicative of better or worse physical health, respectively.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 48
score on a scale | 17.2 [8.1 to 26.9] | 15.9 [10.4 to 22.8]

9. Other Pre Specified Outcome: Health-related Quality of Life, Short Form-36 Mental Component Score
Description: The Short Form-36 (SF-36) mental component score (MCS) was calculated after 6 months of intensive dietetic advice and nutritional support according to well-defined guidelines as follows: 1) recoding of 10 questions of the SF-36 survey; 2) calculation of raw scores for each of the eight health state domains of the SF-36 survey; 3) transformation of raw scores into a 0-100 scale; 4) standardisation of the transformed scales using a z-score transformation and the means and standard deviations from the general United Kingdom (UK) population; 5) calculation of the MCS by multiplying each scale z-score by their respective mental factor score coefficient and summing the eight products; and 6) the resulting sum is multiplied by 10 and added to 50 to linearly transform the MCS to the T-score metric, which has a mean of 50 and a standard deviation of 10 for the general UK population. A MCS score above or below 50 is therefore indicative of better or worse mental health, respectively.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 48
score on a scale | 47.5 [38.5 to 57.3] | 41.6 [30.6 to 49.9]

10. Other Pre Specified Outcome: Health-related Quality of Life, European QoL-5 Dimensions (EQ5D) Health State Score (HSS)
Description: EQ5D HSS after 6 months of intensive dietetic advice and nutritional support. The HSS ranges from -0.285 (for the worst health state) to 1 (for the best health state).
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 48
score on a scale | 0.485 [0.297 to 0.741] | 0.470 [0.198 to 0.699]

11. Other Pre Specified Outcome: Health-related Quality of Life, European QoL-5 Dimensions (EQ5D) Visual Analogue Score (VAS)
Description: EQ5D VAS after 6 months of intensive dietetic advice and support. The VAS uses a thermometer-like scale numbered from 0 to 100 to grade the current health status of individuals; the higher the VAS the better the health state.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 28 | 48
score on a scale | 45 [27 to 60] | 50 [25 to 69]

12. Other Pre Specified Outcome: Deaths/All-cause Mortality
Description: The total number of deaths during follow up was recorded at 6 months.
Time Frame: 6 months
Population: A total of 32 dialysis patients were enrolled at baseline in Study 2. Four patients did not complete the study protocol. Twenty eight patients completed 6 months of intervention and were therefore included in the final analysis. Historical controls were selected from a previous cohort of 151 dialysis patients. Of these, 56 were classified as being malnourished at baseline. Forty nine patients completed 6 months of follow-up and were included in the final analysis.
Measure: Number; unit: participants
Arm/Group | Study 2 - Non Randomised Proof of Principle Study | Historical Control Group From Study 1
Number analyzed (Participants) | 32 | 56
participants | 3 | 5

ADVERSE EVENTS:
Time Frame: The occurrence of an adverse event as a result of participation within this study was not expected and as such no adverse event data was collected.
Description: The occurrence of an adverse event as a result of participation within this study was not expected and as such no adverse event data was collected.
Groups:
- Study 2: Malnourished participants receiving dialysis.
- Historical Control Group: Historical control group of malnourished participants on dialysis taken from Study 1.
Arm/Group | Study 2 | Historical Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This was a single-centre proof of principle study. The number of participants was small and the follow-up period was relatively short. The results observed in this study may not be applicable to populations with dark skin colour (who were excluded from our study) because skin autofluorescence measurements cannot be performed in persons with darker skin colour because of the high absorption of the excitation light.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT02878317/Prot_SAP_000.pdf